CLINICAL TRIAL: NCT06650839
Title: Proof of Concept Clinical Investigation for the Treatment of Subjects With Moderate Aortic Valve Stenosis Using Valvosoft® Non-Invasive Ultrasound Therapy
Brief Title: POC for the Treatment of Subjects With Moderate AS Using Valvosoft® Non-Invasive Ultrasound Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company decision not to start the study
Sponsor: Cardiawave SA (Industry)
Collaborators: Micro Cro (Unknown); TWrite (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW23-02
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Moderate Aortic Valve Stenosis
Keywords: aortic stenosis; moderate; aortic valve; balloon valvuloplasty; TAVR; SAVR; Ultrasound; FUS; PCUT; NIUT
MeSH Terms: conditions — Aortic Valve Stenosis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment MAS (Experimental): Subjects will be treated with Valvosoft, Ultrasound guided Non-Invasive Ultrasound Therapy (NIUT) medical device, to reduce the symptoms caused by moderate aortic stenosis
  Interventions: Device: NIUT

INTERVENTIONS:
Device: NIUT — Treatment of moderate aortic stenosis using non-invasive ultrasound therapy delivered by Valvosoft

SUMMARY:
This study is a proof of concept looking at the safety of treating subjects with moderate aortic stenosis using a Non-Invasive Ultrasound Therapy.

DETAILED DESCRIPTION:
Valvosoft, Ultrasound guided Non-Invasive Ultrasound Therapy (NIUT) medical device, delivers focused and controlled, short ultrasound pulses (<20μsec), directed trans-thoracically at a high acoustic intensity (measured in watts per square centimeter (W/cm2), to produce non-thermal mechanical tissue softening of the targeted calcified aortic valve.

Echocardiographic live imaging enables to follow valve movements in real-time and thus target the therapeutic ultrasound on the calcified valve with great precision. This is first in human or proof of concept study.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic Valve Area (AVA) ≥1.0 cm2 ≤ 1.5 cm2 and either mean aortic Pressure Gradient (mPG) of >25 - < 40 mmHg or maximum velocity (Vmax) ≥3 ≤4 m/sec in normal flow conditions; or
2. Normal-flow, low-gradient aortic stenosis (AS) with preserved ejection fraction (mean aortic Pressure Gradient (mPG) <40 mmHg, Aortic Valve Area (AVA) ≥0.8 ≤1.0 cm2, Left Ventricular Ejection Fraction (LVEF) ≥50%, Stroke Volume Index (SVi) >35 mL/m2);
3. Age ≥18 years;

Exclusion Criteria:

1. mPG ≥40 mmHg; or
2. Severe aortic valve stenosis or other severe valve diseases; or
3. Subject with severe aortic regurgitation; or
4. Subjects with implanted mechanical or bioprosthetic valve in aortic position, or mechanical valve in any other positions; or
5. Heart failure with a NYHA 3 or 4; or
6. Cardiogenic shock or other hemodynamic instability; or
7. LVEF ≤50%; or
8. History of heart transplant; or
9. Subject with a significant kidney disease (eGFR ≤30 mL/min/1.73 m2) or subject is on dialysis; or
10. Subject with uncontrolled hypertension defined as systolic Blood Pressure (BP) ≥160 mmHg and/or a diastolic BP ≥100 mmHg (mean of 3 measurements for both assessments); or
11. Cardiac imaging evidence of vegetation; or
12. Current endocarditis; or 13 Subject has a documented history of cardiac amyloidosis; or

14. Acute Myocardial Infarction (MI) ≤1 month prior to enrolment; or 15. Stroke or Transient Ischemic attack (TIA) ≤1 month prior to enrollment; or 16. Balloon Aortic Valvuloplasty (BAV) ≤3 months prior to enrollment; or 17. Leukopenia (WBC <4000 cell/μL), anemia (Hgb < 8 g/dL), thrombocytopenia (platelet count <50.000 cell/μL), or history of coagulopathy or hypercoagulable state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of MACE | from baseline to 30 days FU
  Rate of MACE defined as a composite of all-cause mortality, MI, stroke, rehospitalization for heart failure at 30 days.
Improvement in leaflet mobility | at 6 months FU compared to baseline
  Change in leaflet mobility measured by means of a change in AVA

SECONDARY OUTCOMES:
Rate of MACE | at 6 , 12 , 18 , 24 months
  Rate of MACE
Rate of all Serious Adverse Events | peri-procedural and at 30 days, 3 , 6 , 12 , 18 , 24 months
  Rate of all Serious Adverse Events
Rate of Stroke | at 30 days, 3 , 6 , 12 , 18 , 24 months
  Rate of stroke (disabling and non-disabling; ischemic and hemorrhagic
Change of AS | at 30 days, 3 , 6 , 12 , 18 , 24 months compared to Baseline;
  Change of AS by means of AVA( assessed by an independent echocardiographic CoreLab
Change in Quality of Life by means of KCCQ | at 30 days, 3 , 6 , 12 , 18 , 24 months compared to Baseline;
  Improvement of quality of life by means of ansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ is a 23-item, self-administered questionnaire.
Change in Quality of Life by means of EQ-5D | at 30 days, 3 , 6 , 12 , 18 , 24 months compared to Baseline;
  Improvement of quality of life by means of EQ-5D. The EQ-5D descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in Exercise capacity | at 30 days, 6 , 12 , 18 , 24 months compared to Baseline;
  Improvement in VO2-max measured during Echo Spiro-Ergometry (ESE)

CONTACTS AND LOCATIONS:
Overall Officials: Milos Velinovic, MD, PhD, Principal Investigator — University Clinical Centre Serbia; Danijela Trifunovic-Zamklar, MD, PhD, Principal Investigator — University Clinical Centre Serbia
Locations (1):
- University Clinical Centre Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No